CLINICAL TRIAL: NCT06195137
Title: Efficacy of Caffeine vs. Alpha-Lipoic Acid in Burning Mouth Syndrome Treatment
Brief Title: Caffeine vs. ALA in BMS Treatment. (BMS: Burning Mouth Syndrome. ALA: Alpha-Lipoic Acid.)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lu Jiang (Other)
Responsible Party: Sponsor-Investigator, Lu Jiang, Clinical Professor, Sichuan University
Organization: Sichuan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCHSIRB-D-2021-407
Record Dates: First submitted 2023-12-03; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Caffeine; Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Caffeine; Thioctic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeine group (Experimental): Burning mouth syndrome (BMS) patients in Caffeine group were provided with BMS disease explanation and psychological counseling. Then they were told to drink instant coffee containing 120-150 mg of the active ingredient caffeine (2 bags of Nescafe Black Coffee, 1.8g each) at a certain point in time from 8:00 to 12:00 every day, for 2 consecutive weeks.
  Interventions: Dietary Supplement: Caffeine
- Alpha Lipoic Acid (ALA) group (Active Comparator): Burning mouth syndrome (BMS) patients in the ALA group were provided with BMS disease explanation and psychological counseling. Then they took α-lipoic acid (ALA) 3 times a day, after meals, 200 mg each time, for 2 consecutive weeks.
  Interventions: Drug: Alpha Lipoic Acid
- Control gruop (No Intervention): Without intervention treatment, we provided BMS patients in Control group with disease explanation and psychological counseling for patients.

INTERVENTIONS:
Dietary Supplement: Caffeine — caffeine supplementation
  Arms: Caffeine group
Drug: Alpha Lipoic Acid — 600-800 mg ALA
  Other Names: ALA
  Arms: Alpha Lipoic Acid (ALA) group

SUMMARY:
The aim of this study was to evaluate the efficacy of caffeine and alpha-lipoic acid in the treatment of burning mouth syndrome by symptom assessment with visual analogue scale.

DETAILED DESCRIPTION:
The etiology of BMS is multifactorial, involving a complex interplay of neuropathic, psychological, neuroendocrine, and immunological factors. Neurologically, BMS has been categorized into three subtypes: peripheral small fiber neuropathy, subclinical trigeminal neuropathy, and inhibitory dopaminergic deficiency. Neuroimaging and peripheral nerve studies have further implicated altered brain activation patterns and increased expression of specific receptors like TRPV1 and P2X3 in the pathogenesis of BMS. Hormonal imbalances, particularly in estrogen levels, have also been suggested to contribute to contribute to the condition.

Caffeine, a xanthine alkaloid chemically known as 1,3,7-trimethylxanthine, is recognized for its diverse biological functions. As a central nervous system stimulant, its primary mechanism involves antagonizing adenosine receptors, thereby enhancing the release of neurotransmitters such as dopamine and norepinephrine, which are known to play roles in analgesic pathways. Caffeine is also noted for its neuroprotective properties and is theorized to reduce the risk of neurodegenerative diseases. It affects the central processing of pain and is involved in regulating circadian rhythms and sleep-wake cycles. Additionally, caffeine has mild anti-inflammatory properties. Its stimulatory effects may also improve mood and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Diagnosis of BMS according to the 3rd edition of the International Classification of Headache Disorders (ICHD-3)
* Daily intraoral burning or dysaesthesia lasting for more than 2 hours for over 3 months
* Normal oral mucosa and sensory testing
* Condition not better accounted for by another ICHD-3 diagnosis

Exclusion Criteria:

1. Secondary BMS due to local or systemic disorders
2. Prior treatment for BMS
3. Psychiatric or progressive neurological disorders
4. Systemic disorders potentially associated with oral disease
5. Long-term history of smoking, drinking, or medication use
6. Consumption of caffeinated products
7. Poor oral hygiene
8. Abnormal blood test results (including blood count, glucose, serum iron, ferritin and transferrin, folic acid, or vitamin B12 levels)
9. Incomplete medical records
10. Unwillingness to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline and 2 weeks after intervention or observation
  During the interview or telephone follow-up with the patient, ask the patient to fill in the VAS rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Jiang, Study Director — Sichuan University
Locations (1):
- West China Hospital of Stomatology, Sichuan University, Chengdu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu C, Yuan P, Qiu X, Liu D, Xu Y, Xiao Y, Zhou S, Zhang Z, Cai S, Ding W, Xu X, Hou F, Jiang L. Short-Term Dietary Caffeine Intake for Alleviating Symptoms of Burning Mouth Syndrome: A Randomised Controlled Comparison With Alpha-Lipoic Acid. J Oral Rehabil. 2025 Jul;52(7):969-978. doi: 10.1111/joor.13957. Epub 2025 Mar 14. PMID 40084800